CLINICAL TRIAL: NCT03547089
Title: A Prospective Trial to Assess Breast Cancer Survivors and Vaginal Atrophy Treatment
Brief Title: A Prospective Trial to Assess Breast Cancer Survivors and Vaginal Atrophy Treatment Outcomes
Acronym: BRAVO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: W. Grant Stevens, MD (Other)
Responsible Party: Sponsor-Investigator, W. Grant Stevens, MD, Director, Marina Plastic Surgery
Organization: Marina Plastic Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI-ISRP-026
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Vaginal Atrophy; Genitourinary System; Disorder, Female; Vaginal Abnormality; Sexual Dysfunction; Sexual Problem
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Viveve treatment (Experimental): Group of women who receive Viveve treatment
  Interventions: Device: Viveve®

INTERVENTIONS:
Device: Viveve® — A single treatment using Viveve® with 110 pulses administered to the vaginal introitus at 90 J/cm2

SUMMARY:
The focus of this study is to assess breast cancer survivors perspectives of Viveve® Treatment using patient reported outcome tools with a focus on symptoms associated with vulvovaginal atrophy/genitourinary syndrome of menopause (GSM). This will be assessed by the FSFI, FSDS-R and DIVA questionnaires.

DETAILED DESCRIPTION:
Breast cancers that are hormone sensitive require estrogen suppression as a part of multimodal treatment. Estrogen suppression also reduces the likelihood of a breast cancer recurrence. Therefore, breast cancer survivors with estrogen sensitive tumors are placed on hormone suppression therapy with either selective estrogen receptor modulators like tamoxifen or aromatase inhibitors like anastrazole. This therapy typically is administered for five years after a cancer diagnosis. Regardless of age or pre-existing menopausal status, the hormone suppression reduces estrogen levels and can either exacerbate existing menopausal symptoms or induce medical menopause in otherwise premenopausal women. This study will evaluate the patient's perspective of vaginal therapy using the Viveve® device in breast cancer patients.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years or older
* Breast cancer survivors defined as women with a history of hormone sensitive breast cancer on tamoxifen
* Self-reported vaginal laxity
* Meet diagnosis of sexual dysfunction
* Patients must be able to understand and willing to sign a written informed consent document and be willing to complete the patient reported outcome tools at the scheduled time points

Exclusion Criteria:

* Cognitive impairment
* Women currently on chemotherapy and/or radiation or who have had their last chemotherapy within 6 months of the intervention
* Women with active breast cancer disease
* Women currently on hormone therapy or who are pregnant
* Women who have had vaginal or pelvic surgery involving the genitalia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Sexual dysfunction | Baseline, 1 month, 3 months, 6 months
  Measurement of changes in sexual dysfunction using the Female Sexual Function Index (FSFI)

SECONDARY OUTCOMES:
Sexual distress | Baseline, 1 month, 3 months, 6 months
  Measurement of changes in sexual distress using the Female Sexual Distress Scale-Revised (FSDS-R)
Vaginal symptoms | Baseline, 1 month, 3 months, 6 months
  Measurement of changes in vaginal symptoms using the Day-to-Day Impact of Vaginal Aging (DIVA) Questionnaire
Vaginal laxity | Baseline, 1 month, 3 months, 6 months
  Measurement of changes in vaginal laxity using the Vaginal Laxity Questionnaire (VLQ)

CONTACTS AND LOCATIONS:
Overall Officials: W G Stevens, MD, Principal Investigator — Marina Plastic Surgery; Ali A Qureshi, MD, Study Director — Marina Plastic Surgery
Locations (1):
- Marina Plastic Surgery Associates, Marina del Rey, California, United States

IPD SHARING:
Plan to Share IPD: Undecided